CLINICAL TRIAL: NCT05501548
Title: Phase II Study of PARP Inhibitor Olaparib and IV Ascorbate in Castration Resistant Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated by the IRB due to low accrual,
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: AstraZeneca (Industry); McGuff Pharmaceuticals, Inc. (Industry); The Marcus Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J21127; IRB00292465 (Other: JHM IRB); ESR 19-20448 (Other: AstraZeneca)
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer; Castration-resistant Prostate Cancer
Keywords: olaparib; ascorbic acid; PARP; PARP-inhibitor
MeSH Terms: conditions — Prostatic Neoplasms | interventions — olaparib; Ascorbic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Olaparib and Vitamin C (Experimental): Olaparib will be administered at 300 mg by mouth, twice daily; ascorbate will be administered at 1 g/kg IV twice weekly at least 24 hours apart, until objective disease progression or unacceptable toxicities or patient withdrawal for other reasons.
  Interventions: Drug: Olaparib; Dietary Supplement: Vitamin C

INTERVENTIONS:
Drug: Olaparib — Olaparib 300mg by mouth twice daily
  Other Names: Lynparza; AZD2281; KU-0059436
Dietary Supplement: Vitamin C — Ascorbic acid 1g/kg administered intravenously twice weekly
  Other Names: Ascorbic acid; L-ascorbic acid; Ascor; A11GA01

SUMMARY:
This is a study to evaluate the safety and clinical activity of the combination of olaparib and high-dose IV ascorbate, as second or later line of therapy, in castration resistant prostate cancer patients with no known DNA repair gene mutations (DDRm). In brief, the primary endpoint is PSA50 response , defined by a 50% reduction in PSA from baseline . The secondary endpoints are assessing the PSA doubling time, radiographic and PSA PFS, safety and tolerability as defined by the incidence of grade 3 to 5 toxicities, and measuring overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Have metastatic castration-resistant prostate cancer (prostate cancer progressing by PSA (rise by 25% on prior therapy) or imaging despite castrate levels of testosterone [<50 ng/dL] using standard measures of progression defined by Prostate Cancer Working Group3)
* Have a minimum PSA of 1 ng/mL
* Have a pathological diagnosis of prostate carcinoma
* Patients should continue receiving continuous hormonal ablation with surgical or medical castration with baseline testosterone <50ng/dL
* Patients may be receiving bone-targeted agents
* May have received multiple lines of therapy including radium 223, sipuleucel T, and up to 2 lines of chemotherapy (One of 2 lines may be for hormone sensitive metastatic prostate cancer or both can be for castration resistant).
* Age >= 18
* Have ECOG performance status 0-1 (Appendix A)
* Be able to take oral medication and willing to consider a port for ease of administration of ascorbate
* Must have progressed on one systemic line of treatment (can include LHRH agonist/antagonist or orchiectomy and one additional line of therapy (abiraterone, enzalutamide, apalutamide, darolutamide, docetaxel, etc))
* Have normal organ and marrow function measured within 28 days prior to administration of study treatment as defined below:

  * Absolute neutrophil count >1.5 x 109/L
  * Platelets ≥ 100,000/mm³
  * Hemoglobin ≥ 9g/dL with no blood transfusion in the past 28 days
  * Total bilirubin ≤ 1.5 ULN
  * AST (SGOT)/ALT(SGPT) ≤ 2.5 x ULN (≤5x ULN if with known liver metastases provided bilirubin is normal
  * Creatinine ≤ 1.6 x ULN (for patients with ≥1.6 x ULN, calculated or measured creatinine clearance must be ≥ 60 mL/minute (Cockcroft-Gault)
* Men of reproductive potential and those who are surgically sterilized (i.e. post- vasectomy) must agree to practice effective barrier contraception that has an expected failure rate of <1% during and for 6 months after discontinuation of study treatment. Female partners should also use a highly effective form of contraception ([see Appendix C for acceptable methods]) if they are of childbearing potential.

  * If condoms are used as a barrier contraceptive, a spermicidal agent should be added to ensure that pregnancy does not occur
* Have the ability to understand, and have given written informed consent before performance of any study-related procedures not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

* Have a known DNA repair mutation (minimum list of genes that must be mutation negative for inclusion: ATM, BARD1, BRCA1, BRCA2, BRIP1, CDK12, CHEK1, CHEK2, FANCL, PALB2, RAD51B, RAD51C, RAD51D, RAD45L). In addition, patients who have not completed germline and somatic testing to rule out such a mutation are ineligible until they have completed testing. If tissue or liquid ctDNA sequencing was not previously done, testing using the Foundation One liquid biopsy test or an equivalent FDA-approved test is acceptable as standard of care.

  * DNA repair mutation variant of unknown significance (VUS) allowed
* Have had known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
* No prior olaparib, rucaparib, or other PARP inhibitor
* Have had major surgery within 2 weeks of dosing of investigational agent
* Have had palliative radiation or another biological cancer therapy within 2 weeks prior to the first dose of study drug (2 week wash out required)
* Patients receiving any systemic chemotherapy or radiotherapy within 3 weeks prior to study treatment
* Have received other investigational drugs within 14 days prior to enrollment.
* Is expected to require chemotherapy or radiation for pain palliation in the next 12 weeks.
* Have used or plan concomitant use of the following medications in the past 6 months prior to enrollment: 5-alpha reductase inhibitors unless subject has been taking stable dose of medication for prior 6 months
* Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study treatment is 2 weeks. See the following link for a complete list of known CYP3A inhibitors: https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers
* Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents. See the following link for a complete list of known CYP3A inhibitors:https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers
* Have moderate or severe cardiovascular disease:

  * Has the presence of cardiac disease, including a myocardial infarction within six months prior to study entry, unstable angina pectoris, New York Heart Association Class III/IV congestive heart failure, or uncontrolled hypertension.
  * Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (eg., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTc prolongation >500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
* Have uncontrolled intercurrent illness, including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Other malignancy unless curatively treated with no evidence of disease for >5 years except adequately treated non-melanoma skin cancer
* Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia
* Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Patients with known active hepatitis (i.e. Hepatitis B or C)
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Channing Paller, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Olaparib and Vitamin C
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Olaparib and Vitamin C
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: PSA50 Response
Description: Number of participants with metastatic castration resistance prostate cancer (mCRPC) who experience a 50% reduction in prostate specific antigen (PSA50) from baseline. PSA50 response will be defined as a decrease in the PSA to 50% less than the baseline PSA upon enrollment in the trial. The decrease must be confirmed by a second measurement at least 4 weeks apart. PSA values will be measured monthly during the trial.
Time Frame: up to 5 years
Population: Data was not collected for this outcome measure.
Arm/Group | Olaparib and Vitamin C
Number analyzed (Participants) | 0

2. Secondary Outcome: Safety and Tolerability of Olaparib in Combination With IV Ascorbic Acid in Patients With mCRPC
Description: Number of participants experiencing treatment-related adverse events as defined by NCI CTCAE v5.0.
Time Frame: up to 1 year 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib and Vitamin C
Number analyzed (Participants) | 4
Participants | 4

3. Secondary Outcome: PSA Doubling Time in Patients With mCRPC Receiving Olaparib in Combination With IV Ascorbic Acid
Description: Median number of months to PSA doubling from the initiation of therapy until the PSA has increased to 200% of baseline value, and confirmed with another measurement at least 4 weeks later, or death. The date of PSA doubling will be the first value recorded (not the confirmatory value).
Time Frame: up to 5 years
Population: Data was not collected for this outcome measure.
Arm/Group | Olaparib and Vitamin C
Number analyzed (Participants) | 0

4. Secondary Outcome: Radiographic Progression Free Survival (rPFS) of Patients With mCRPC Receiving Olaparib in Combination With IV Ascorbic Acid
Description: Number of months from initiation of therapy to date of first radiographic progression, death from any cause, or last patient evaluation. Radiographic progression will be defined as soft tissue disease progression by modified RECIST criteria 1.1 (baseline LN size must be >1.0 cm to be considered target or evaluable lesion) or by development of two or more new bone lesions not consistent with tumor flair for prostate cancer working group 3.
Time Frame: up to 5 years
Population: Data was not collected for this outcome measure.
Arm/Group | Olaparib and Vitamin C
Number analyzed (Participants) | 0

5. Secondary Outcome: PSA Progression Free Survival (PSA PFS) of Patients With mCRPC Receiving Olaparib in Combination With IV Ascorbic Acid
Description: Number of months to first PSA failure (two consecutive increases in PSA of 50% and >=5ng/mL above nadir) or death
Time Frame: up to 5 years
Population: Data was not collected for this outcome measure.
Arm/Group | Olaparib and Vitamin C
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival of Patients With mCRPC Receiving Olaparib in Combination With IV Ascorbic Acid
Description: Number of months from initiation of therapy to death due to any cause
Time Frame: up to 5 years
Population: Data was not collected for this outcome measure.
Arm/Group | Olaparib and Vitamin C
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From enrollment through study completion (approximately 1 year 4 months)
Arm/Group | Olaparib and Vitamin C
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib and Vitamin C (N=4)
Headache (Nervous system disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Dry eye (Eye disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Chills (General disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 4 (4)
Flushing (Vascular disorders) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Pain (General disorders) | 2 (3)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT05501548/Prot_SAP_000.pdf